CLINICAL TRIAL: NCT03760159
Title: Minimally Invasive Detection of a Sleep Apnoea and Effects of nCPAP Therapy : a Proof-of-concept Study
Brief Title: Minimally Invasive Detection of a Sleep Apnoea
Acronym: KCG_SLEEP
Status: Terminated | Type: Observational
Why Stopped: Terminated because sample size achieved
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2018/290
Record Dates: First submitted 2018-10-19; First posted 2018-11-30 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Sleep Disorder; Breathing-Related; Cardiovascular Diseases; Cardiovascular Risk Factor; Cardiovascular Complication
MeSH Terms: conditions — Sleep Wake Disorders; Cardiovascular Diseases | interventions — Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group RESPIRATORY SIMUL (Study A): In 46 healthy subjects, a computer program will generate random instructions of periods of normal breathing, voluntary end-expiratory breathing cessation periods (as surrogate of central apnoea) and Muller's manœuvre (as surrogate of obstructive apnoea). Meanwhile, the KCG will record the parameters of biological interest. ECG, heart rate, beat to beat non-invasive blood pressure (Finometer), ventilation, end-tidal CO2 (AD instruments), O2 saturation (Nellcor), cardiac output (CO) (Philips) will also be recorded.
  Interventions: Device: Kinocardiography unintrusive recording
- Group SDB (Study B): In patients suspected of sleep apnoea and admitted to the sleep unit of the Erasme hospital to perform sleep test as required by their medical condition, the investigators will simultaneously record KCG and PSG and qualitatively compare the data (Bland-Altman plots).
  Interventions: Device: Kinocardiography unintrusive recording
- Group nCPAP (Study C): In patients with a diagnosis of sleep apnea, the investigators will determine if KCG is capable to reliably assess the efficacy of the nCPAP therapy in comparison to simultaneous PSG recording. Ongoing adjustment in the CPAP therapy pressure during the night, and its effect on cardiovascular haemodynamic assessed by the KCG, will be taken into account as well.
  Interventions: Device: Kinocardiography unintrusive recording
- Group UNSELECTED (Study D): After validation of the three previous steps, the investigators plan to extend the recordings on 100 unselected consecutive patients, without recruitment restrictions, which will undergo PSG recordings because of complains of sleep apnoea.
  Interventions: Device: Kinocardiography unintrusive recording

INTERVENTIONS:
Device: Kinocardiography unintrusive recording — The Kinocardiography (Kino) is a device which records the electric and mechanic function of the heart. The device comprises a combination of ECG recording, (6 degrees of freedom), accelerometer and gyroscope sensors. The Kino device consists of a back and a chest housing in contact with the patient. The back housing is placed in the middle of the lower back of the patient, and the chest housing is placed on the chest (either on the sternum or on the costal grill at the apex of the heart). The housings are connected by two cables. Data obtained from the device are visualized on a digital application via a Bluetooth connection.
  For the group A, the KCG records the cardiac signals while the patient performs specific respiratory manoevres, as describe above.
  For group B, C, D, the KCG records the cardiac contraction during sleep along with the PSG recording.
  Other Names: For Group A, recording of the follow: heart rate, humeral blood pressure, oxygen saturation, respiratory rate, cutaneous pO2, pCO2, endtidalCO2,

SUMMARY:
Obstructive sleep apnoea (OSA) is characterised by recurrent nocturnal respiratory interruptions, resulting from the total or partial collapse of the upper respiratory ways. This results into sleep fragmentation, metabolic and biological disorders, which alter the neuropsychological and cardiovascular systems. Nowadays, 24% of men and 9% of women aged 30 to 60 years disclose already an asymptomatic and underdiagnosed sleep disorder breathing (SDB). In subjects suffering from cardiovascular disease, prevalence of SDB is higher than in the general population, reaching 87% in people with resistant hypertension, 51% in those with heart failure and 62% in those with atrial fibrillation (to cite a few).The current diagnostic tool for SDB is polysomnography (PSG), but this is an expensive, time-consuming and uncomfortable tool, which limits its wide-spread use despite the high frequency of SDB in general and, even more, in patients suffering from cardiovascular diseases. Several screening devices exist in order to test those patients at risk of SDB, but these have several limitations, since they are not recommended in patients who are asymptomatic for apnoea, in those with cardiorespiratory diseases, nocturnal arrhythmias or neurological and metabolic co-morbidities. In other words, nowadays there isn't an efficient screening tool of SDB, mainly for those with a low pre-test probability of having SDB.

Preliminary evidence suggests that the seismocardiography (SCG) and the ballistocardiography (BCG) can detect nocturnal awakening and sleep disturbances with a good sensitivity and accuracy as compared to the state-of-the-art PSG. Simultaneous recording of SCG and BCG is called kinocardiography (KCG) and has not been performed yet during sleep.

The main hypothesis tested in this study is that the KCG provides sensitive and accurate measures of obstructive and central apnoea as compared to the state-of-the-art PSG. The secondary hypotheses are related to modifications in the SCG and BCG signals during the apnoea and the effects of continuous positive air pressure (CPAP) therapy. These hypotheses will be tested through a series of studies in normal volunteers and patients, as follow:

* Group RESPIRATOIRYSIMUL (Study A): voluntary end-expiratory breathing cessations periods and obstructive voluntary apnoea's (n=46);
* Group SBD (Study B): patients admitted for complains of sleep disturbances without cardiovascular and/or respiratory abnormalities which could induce artifacts in the KCG recording (n=50);
* Group nCPAP (Study C): patients treated by nCPAP therapy (n=50);
* Group UNSELECTED (Study D): unselected consecutive patients (n=100), without recruitment restrictions.

Study A is an interventional study on voluntary breath holding in normal volunteers. Studies B, C and D are observational investigations recruiting subjects referred for PSG as required by their medical condition. Because the KCG device is not intrusive, the investigators do not anticipate difficulties in the enrollment. This study will not affect in any manner the regular medical care of the patients admitted to the sleep laboratory.

To conclude, SDB is a widespread disease with detrimental health effects and its prevalence is supposed to increase in future years. PSG is the gold standard for diagnosis of SDB but it is an expensive, uncomfortable and time-consuming tool, limiting its use in daily clinical practice. For subjects with a high pre-test probability of SDB, portable, inexpensive and easy-to-use tools have been proposed as sleep monitoring and seem to provide accurate estimates of SDB. Although such devices seem promising, they disclose also several limitations and are not universally accepted as SDB screening devices, mainly in case of low pre-test probability of SBD. The less cumbersome KCG may screen patients for SDB accurately. One of its unique features is also that it can directly identify the consequences of SDB and nCPAP therapy on the cardiovascular system, and in especially the presence of frequently associated cardiac arrhythmias. With a more efficient pre-screening, those who are most likely to be eligible for nCPAP therapy will have a better access to the currently existing sleep laboratory facilities. The present research project has thus the potential of improving SDB patients care and health, at no additional societal costs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-70 years old

Exclusion Criteria (group A):

* Cardiorespiratory co-morbidities

Exclusion Criteria (groups B-C-D):

* BMI>35 kg/m2
* Moderate, severe valvular disease
* Permanent atrial fibrillation or frequent premature contractions
* Atrio-ventricular conduction disturbances
* Medications which reduces heart rate and heart rate variability
* Cardiac rhythm driven by a pacemaker
* Systolic heart failure of any origin (ischaemic, dilatated ect..)
* Neurological diseases responsible for abnormal movements
* Denied participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A includes health voluntary subject, without cardiorespiratory co-morbidities.
  Groups B and C include patients admitted to the sleep laboratory to perform a PSG because of clinical suspicion of SDB.
  Group D includes 100 unselected consecutive patients who will undergo PSG recordings because of complains of sleep apnoea.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Group RESPIRATORY SIMUL (Study A) | Three months
  The BCG and SCG kinetic energy (mJ) recorded with the KCG are profoundly affected by abnormal respiration, mainly by the Muller's manoeuvre.
Group RESPIRATORY SIMUL (Study A) | Three months
  The BCG and SCG kinetic energy changes are correlected with the changes of the intrathoracic pressure
Group SDB (Study B) | One year
  The BCG and SCG signals are profoundly affected by the apnoea itself. The magnitude of these changes dépends on the severity of the underlying apnoea itself.
Group nCPAP (Study C) | One year
  The BCG and SCG signals are reversed to the Baseline in patients treated with nCPAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Morra, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morra S, Hossein A, Gorlier D, Rabineau J, Chaumont M, Migeotte PF, van de Borne P. Modification of the mechanical cardiac performance during end-expiratory voluntary apnea recorded with ballistocardiography and seismocardiography. Physiol Meas. 2019 Nov 4;40(10):105005. doi: 10.1088/1361-6579/ab4a6a. PMID 31579047

DOCUMENTS (1):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03760159/Prot_000.pdf